CLINICAL TRIAL: NCT02563314
Title: Comparison of Two Oxygen Setting During Non-invasive Mechanical Ventilation of Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Comparison of Two Oxygen Setting During Non-invasive Mechanical Ventilation of Chronic Obstructive Pulmonary Disease
Acronym: OXYSET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of the coordinating investigator from another institution
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1408025; ANSM (Other: 2014-A00319-38)
Record Dates: First submitted 2015-09-24; First posted 2015-09-30 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease With Acute Exacerbation, Unspecified
Keywords: Noninvasive Ventilation; Pulmonary Disease; Chronic Obstructive; Renal Doppler; Oxygen; Hypercapnia
MeSH Terms: conditions — Lung Diseases; Hypercapnia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Device: Non-invasive mechanical ventilation - Normoxia
- control (Other)
  Interventions: Device: Non-invasive mechanical ventilation - Controlled hypoxemia

INTERVENTIONS:
Device: Non-invasive mechanical ventilation - Normoxia — Maintenance of an oxygen setting allowing normal oxygen saturation during non-invasive mechanical ventilation (SpO2 targeted 96-98%)
  Arms: intervention
Device: Non-invasive mechanical ventilation - Controlled hypoxemia — Maintenance of an oxygen setting allowing mild hypoxemia during non-invasive mechanical ventilation (SpO2 targeted 88-92%)
  Arms: control

SUMMARY:
Hypoxaemic patients with exacerbations of chronic obstructive pulmonary disease (COPD) are at some risk of carbon dioxide (CO2) retention during oxygen therapy. Main mechanism of CO2 retention is believed to be reversal of preexisting regional hypoxic pulmonary vasoconstriction, resulting in a greater dead space. Risk of CO2 retention during mechanical ventilation remains controversial. Thus recent study suggested limited risk of CO2 retention with controlled oxygen supplementation during mechanical ventilation. Conversely, controlled oxygen supplementation might decrease dyspnea and respiratory workload, increase comfort and improve both urinary output and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute hypercapnic COPD exacerbation
* Respiratory acidosis
* Intensive care unit admission
* Non-Invasive mechanical ventilation for less than 24 hours
* Patients or proxy consent
* Patients affiliated with the General Social Security Health System

Exclusion Criteria:

* Pregnancy
* Sickle cells disease
* Acute coronary syndrome
* Restrictive respiratory disease
* Stage 4 or 5 chronic kidney disease
* COPD exacerbation following a first episode of conventional mechanical ventilation
* Contraindications to non-invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
urinary output (ml) | 24 hours
  First 24 hours of non-invasive mechanical ventilation

SECONDARY OUTCOMES:
Changes in CO2 levels | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
respiratory workload during non-invasive mechanical ventilation (occlusion pressure (cm H2O) to 100 ms after the onset of inspiration) | 24 hours, 48 hours, 72 hours
  First 24 hours of non-invasive mechanical ventilation
Serum creatinine | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Renal resistive index | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Pulmonary arterial pressure | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Semiquantitative assessment of dyspnea (visual likert scale) | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Semiquantitative assessment of comfort (visual likert scale) | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Fluid balance | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
SOFA (Sequential Organ Failure Assessment) score | 24 hours, 48 hours, 72hours
  First 24 hours of non-invasive mechanical ventilation
Mortality | up to day 28
  First 24 hours of non-invasive mechanical ventilation
Number of patients requiring mechanical ventilation | up to day 28
  Evaluation until 28 days with an evaluation at intensive care unit discharge, and at hospital discharge
days alive without mechanical ventilation | up to day 28
  Evaluation up to 28 days with an evaluation at intensive care unit discharge, and at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael DARMON, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (4):
- France (4):
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand
  - CHu de GRENOBLE, Grenoble
  - CHU de la Pitié-Salpêtrière, Paris
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No